CLINICAL TRIAL: NCT00630877
Title: A Randomized, Double-blind, Parallel, Multicenter, Placebo-controlled, Prospective Study to Evaluate the Functionality of the Flushing ASsessment Tool (FAST) in Subjects Administered Niaspan® Plus Acetylsalicylic Acid (ASA), Niaspan® Plus ASA Placebo or Niaspan® Placebo Plus ASA Placebo Daily for Six Weeks
Brief Title: Evaluation of a Flushing ASsessment Tool (FAST) in Subjects Receiving Niacin Extended-release Plus Aspirin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Scott Krause, Associate Director, Clinical Research, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-229
Record Dates: First submitted 2008-02-29; First posted 2008-03-07 (Estimated); Results first posted 2009-10-09 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-09

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NER/ASA (Experimental)
  Interventions: Drug: Niacin extended-release (NER); Drug: Aspirin (ASA)
- NER/ASA Placebo (Experimental)
  Interventions: Drug: Niacin extended-release (NER); Drug: Aspirin (ASA) placebo
- NER Placebo/ASA Placebo (Experimental)
  Interventions: Drug: Niacin extended-release (NER) placebo; Drug: Aspirin (ASA) placebo

INTERVENTIONS:
Drug: Niacin extended-release (NER) — Tablets administered once daily for 6 weeks; titrated to a maximum dose of 2000 mg
  Other Names: ABT-919; Niaspan
  Arms: NER/ASA; NER/ASA Placebo
Drug: Niacin extended-release (NER) placebo — Tablets administered once daily for 6 weeks
  Arms: NER Placebo/ASA Placebo
Drug: Aspirin (ASA) — Tablets (325 mg) administered once daily for 6 weeks
  Other Names: acetylsalicylic acid
  Arms: NER/ASA
Drug: Aspirin (ASA) placebo — Tablets administered once daily for 6 weeks
  Arms: NER Placebo/ASA Placebo; NER/ASA Placebo

SUMMARY:
The primary purpose of this study was to evaluate the psychometric characteristics (reliability, validity, and responsiveness) of a Flushing ASsessment Tool (FAST) in subjects receiving niacin extended-release (NER) plus aspirin (ASA) daily for 6 weeks.

The FAST is a questionnaire that was developed to provide a detailed assessment of flushing symptoms and their impact in patients receiving niacin therapy. The effect of aspirin on flushing symptoms, as measured by the FAST, was also evaluated.

DETAILED DESCRIPTION:
This study was designed to evaluate the psychometric characteristics of the FAST questionnaire.

The FAST is a self-administered questionnaire, completed using a hand-held electronic data capture device (LogPad e-diary). Subjects recorded the start and stop date and time of each flushing event, the presence and severity of individual flushing symptoms (redness, warmth, tingling and/or itching), and an overall assessment of their flushing experience.

Evaluation of the psychometric characteristics of the FAST was based on 3 primary data analyses: 1 ) test-retest reliability based on the intraclass correlation coefficient; 2) construct validity based on Spearman correlation coefficients; and 3) responsiveness based on changes in FAST scores. The mean and maximum severity of flushing events, as measured by the FAST, were the primary variables evaluated in each of the 3 data analyses mentioned above. Psychometric analyses were performed blinded to treatment group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least one year or surgically sterile, or is of childbearing potential and must agree to practice birth control for the duration of the study.
* Have dyslipidemia as demonstrated by laboratory results.

Exclusion Criteria:

* Have glycosylated hemoglobin (HbA1c) >= 9.0%.
* Have nephrotic syndrome, dysproteinemias, or severe renal failure (glomerular filtration rate [GFR] < 30 mL/minute, as calculated from creatinine clearance).
* Have had unstable angina or an acute myocardial infarction (MI) within three months of the Screening Visit.
* Have had severe peripheral artery disease as evidenced by intermittent claudication within three months of the Screening Visit.
* Have had uncontrolled cardiac arrhythmias within three months of the Screening Visit.
* Have symptomatic heart failure defined as dyspnea at rest or with exertion (mild peripheral edema is not exclusionary).
* Have a systolic blood pressure measurement of > 180 mmHg or a diastolic blood pressure measurement of > 110 mmHg at the Screening or Baseline Visit
* Have active gout or uric acid >= 11 mg/dL.
* Have a history of hepatitis (acute or chronic), obstructive liver disease, or alanine aminotransferase (ALT; serum glutamic pyruvic transaminase [SGPT]) or aspartate aminotransferase (AST; serum glutamic oxaloacetic transaminase [SGOT]) values >= 1.3 times the upper limit of normal (ULN) at the Screening Visit.
* Have creatine phosphokinase (CPK) >= 3 x ULN at the Screening Visit.
* Have used an investigational study drug or participated in an investigational study within 30 days of the Screening Visit.
* Have a health condition or laboratory abnormality (inclusive of clinically significant laboratory results at Screening Visit), which, in the opinion of the Investigator, may be adversely affected by the procedures or study medications in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Thakkar, MD, Study Director — Abbott
Locations (38):
- United States (38):
  - Birmingham, Alabama
  - Anaheim, California
  - Walnut Creek, California
  - Denver, Colorado
  - Brooksville, Florida
  - Daytona Beach, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Largo, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Arkansas City, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Durham, North Carolina
  - High Point, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greer, South Carolina
  - Austin, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Magna, Utah
  - Murray, Utah
  - Sandy City, Utah
  - Gig Harbor, Washington
  - Menomonee Falls, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Kawata AK, Revicki DA, Thakkar R, Jiang P, Krause S, Davidson MH, Punzi HA, Padley RJ. Flushing ASsessment Tool (FAST): psychometric properties of a new measure assessing flushing symptoms and clinical impact of niacin therapy. Clin Drug Investig. 2009;29(4):215-29. doi: 10.2165/00044011-200929040-00001. PMID 19301936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 41 sites in the United States between February and June, 2008.
Pre-assignment Details: Of the 276 subjects that were randomized, 5 discontinued from the study prior to receiving study drug due to withdrawal of consent (2), death in the family (1), positive pregnancy test (1), and lost to follow up (1).
Groups:
- NER/ASA: Niacin extended-release (NER) titrated to 2000 mg plus aspirin (ASA) 325 mg once daily
- NER/ASA Placebo: Niacin extended-release (NER) titrated to 2000 mg plus aspirin (ASA) placebo once daily
- NER Placebo/ASA Placebo: Niacin extended-release (NER) placebo plus aspirin (ASA) placebo once daily
Period: Overall Study
Arm/Group | NER/ASA | NER/ASA Placebo | NER Placebo/ASA Placebo
Started | 91 (For all arms, started means treated.) | 90 | 90
Completed | 72 | 75 | 80
Not Completed | 19 | 15 | 10
Not completed — Adverse Event | 11 | 8 | 7
Not completed — Withdrawal by Subject | 3 | 4 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Noncompliance | 2 | 3 | 1
Not completed — Protocol violation | 1 | 0 | 1
Not completed — Personal reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NER/ASA | NER/ASA Placebo | NER Placebo/ASA Placebo | Total
Number analyzed (Participants) | 91 | 90 | 90 | 271
Age Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.68) | 53.7 (12.74) | 52.9 (12.26) | 53.6 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 42 | 125
  Male | 49 | 49 | 48 | 146
Region of Enrollment [Number; unit: participants]
  United States | 91 | 90 | 90 | 271

OUTCOME MEASURES:

1. Primary Outcome: Flushing ASsessment Tool (FAST) Test-retest Reliability--mean Flushing Severity Score
Description: Test-retest reliability of the mean flushing severity score was evaluated. The intraclass correlation coefficient comparing flushing severity scores for Week 1 and Week 2 was examined to determine test-retest reliability. Flushing severity was assessed using the FAST on a scale of 1 to 10, with 10 being the most severe.
Time Frame: Week 1 to Week 2
Population: Subjects with stable flushing symptoms from Week 1 to Week 2.
Measure: Number; unit: Intraclass correlation coefficient
Groups:
- Subjects With Stable Flushing Symptoms: Subjects whose flushing symptoms remained stable from Week 1 to Week 2
Arm/Group | Subjects With Stable Flushing Symptoms
Number analyzed (Participants) | 174
Intraclass correlation coefficient | 0.75

2. Secondary Outcome: Maximum Severity of Flushing Events Overall During the Study
Description: The severity of flushing events was assessed as none, mild, moderate, severe, or very severe using the FAST. The maximum severity of flushing events overall during the study was compared among treatment groups.
Time Frame: Week 1 to Week 6
Population: m-ITT population, defined as all randomized subjects who received at least 1 dose of study drug and who had at least 1 entry in the e-diary.
Measure: Number; unit: Percentage of subjects
Arm/Group | NER/ASA | NER/ASA Placebo | NER Placebo/ASA Placebo
Number analyzed (Participants) | 90 | 90 | 89
Percentage of subjects
  None | 26 | 14 | 37
  Mild | 23 | 16 | 38
  None/Mild | 49 | 30 | 75
  Moderate | 34 | 31 | 22
  Severe | 17 | 32 | 2
  Very Severe | 0 | 7 | 0
Statistical Analysis 1: Comparison: NER/ASA vs NER/ASA Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

3. Primary Outcome: FAST Test-retest Reliability--maximum Flushing Severity Score
Description: Test-retest reliability of the maximum flushing severity score was evaluated. The intraclass correlation coefficient comparing flushing severity scores for Week 1 and Week 2 was examined to determine test-retest reliability. Flushing severity was assessed using the FAST on a scale of 1 to 10, with 10 being the most severe.
Time Frame: Week 1 to Week 2
Population: Subjects with stable flushing symptoms from Week 1 to Week 2.
Measure: Number; unit: Intraclass correlation coefficient
Arm/Group | Subjects With Stable Flushing Symptoms
Number analyzed (Participants) | 174
Intraclass correlation coefficient | 0.40

4. Primary Outcome: FAST Cross-sectional Construct Validity--mean Flushing Severity Score
Description: The relationship between mean flushing severity and overall flushing troublesomeness was evaluated by examining the Spearman rank-order correlation. Flushing severity was assessed using the FAST on a scale of 1 to 10, with 10 being the most severe. Overall flushing troublesomeness was assessed using the FAST on a scale of 1 to 10, with 10 being the most troublesome.
Time Frame: Week 1
Population: as for outcome 2
Measure: Number; unit: Spearman correlation coefficient
Groups:
- Modified Intent-to-Treat (m-ITT) Population: All subjects who received study drug and had an entry in the e-diary.
Arm/Group | Modified Intent-to-Treat (m-ITT) Population
Number analyzed (Participants) | 269
Spearman correlation coefficient | 0.64
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (m-ITT) Population; Test type: Superiority or Other; p < 0.0001, Spearman rank-order correlation

5. Primary Outcome: FAST Cross-sectional Construct Validity--maximum Flushing Severity Score
Description: The relationship between maximum flushing severity and overall flushing troublesomeness was evaluated by examining the Spearman rank-order correlation. Flushing severity was assessed using the FAST on a scale of 1 to 10, with 10 being the most severe. Overall flushing troublesomeness was assessed using the FAST on a scale of 1 to 10, with 10 being the most troublesome.
Time Frame: Week 1
Population: as for outcome 2
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Modified Intent-to-Treat (m-ITT) Population
Number analyzed (Participants) | 269
Spearman correlation coefficient | 0.66
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (m-ITT) Population; Test type: Superiority or Other; p < 0.0001, Spearman rank-order correlation

6. Primary Outcome: FAST Longitudinal Construct Validity--mean Flushing Severity Score
Description: The relationship between the change in mean flushing severity scores from Week 1 to Week 2, and the subject-rated overall treatment effect scale administered at Week 2, was assessed by examining the Spearman rank-order correlation. Flushing severity was assessed using the FAST on a scale of 1 to 10, with 10 being the most severe. The overall treatment effect was assessed on a scale of 1 (symptoms are worse since study start), 2 (symptoms are about the same since study start), or 3 (symptoms are better since study start).
Time Frame: Week 1 to Week 2
Population: as for outcome 2
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Modified Intent-to-Treat (m-ITT) Population
Number analyzed (Participants) | 269
Spearman correlation coefficient | -0.44
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (m-ITT) Population; Test type: Superiority or Other; p < 0.0001, Spearman rank-order correlation

7. Primary Outcome: FAST Longitudinal Construct Validity--maximum Flushing Severity Score
Description: The relationship between the change in maximum flushing severity scores from Week 1 to Week 2, and the subject-rated overall treatment effect scale administered at Week 2, was assessed by examining the Spearman rank-order correlation. Flushing severity was assessed using the FAST on a scale of 1 to 10, with 10 being the most severe. The overall treatment effect was assessed on a scale of 1 (symptoms are worse since study start), 2 (symptoms are about the same since study start), or 3 (symptoms are better since study start).
Time Frame: Week 1 to Week 2
Population: as for outcome 2
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Modified Intent-to-Treat (m-ITT) Population
Number analyzed (Participants) | 269
Spearman correlation coefficient | -0.42
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (m-ITT) Population; Test type: Superiority or Other; p < 0.0001, Spearman rank-order correlation

8. Primary Outcome: FAST Responsiveness--mean Flushing Severity Score
Description: The change in mean flushing severity scores from study start to Day 43 was compared in subjects classified as responders vs. nonresponders. Flushing severity was assessed using the FAST on a scale of 1 to 10, with 10 being the most severe. Changes in mean flushing severity scores were negative if flushing symptoms improved and positive if flushing symptoms worsened.
Time Frame: Study start to Day 43
Population: Subjects in the m-ITT population were classified as responders (improved flushing symptoms) or nonresponders (no change or worsened flushing symptoms) based on changes in flushing symptoms from study start to Day 43.
Measure: Number; unit: Units on a scale
Groups:
- Responders: Subjects whose flushing symptoms improved from study start to Day 43.
- Nonresponders: Subjects whose flushing symptoms did not change or worsened from study start to Day 43.
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 46 | 159
Units on a scale | -0.51 | 0.15
Statistical Analysis 1: Comparison: Responders vs Nonresponders; Test type: Superiority or Other; p = 0.002, Independent groups t-test

9. Primary Outcome: FAST Responsiveness--maximum Flushing Severity Score
Description: The change in maximum flushing severity scores from study start to Day 43 was compared in subjects classified as responders vs. nonresponders. Flushing severity was assessed using the FAST on a scale of 1 to 10, with 10 being the most severe. Changes in maximum flushing severity scores were negative if flushing symptoms improved and positive if flushing symptoms worsened.
Time Frame: Study start to Day 43
Population: as for outcome 8
Measure: Number; unit: Units on a scale
Arm/Group | Responders | Nonresponders
Number analyzed (Participants) | 46 | 159
Units on a scale | -1.85 | -0.18
Statistical Analysis 1: Comparison: Responders vs Nonresponders; Test type: Superiority or Other; p < 0.001, Independent groups t-test

ADVERSE EVENTS:
Arm/Group | NER/ASA | NER/ASA Placebo | NER Placebo/ASA Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 1 | 2
Other Adverse Events (participants affected / at risk) | 74 | 80 | 60
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | NER/ASA | NER/ASA Placebo | NER Placebo/ASA Placebo
Non-cardiac chest pain (General disorders) | 1/91 (1) | 0/90 (0) | 0/90 (0)
Myocardial infarction (Cardiac disorders) | 0/91 (0) | 1/90 (1) | 0/90 (0)
Right renal cyst (Renal and urinary disorders) | 0/91 (0) | 0/90 (0) | 1/90 (1)
Nephrolithiasis (Renal and urinary disorders) | 0/91 (0) | 0/90 (0) | 1/90 (1)
Adenomatous polyposis (Congenital, familial and genetic disorders) | 0/91 (0) | 0/90 (0) | 1/90 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | NER/ASA | NER/ASA Placebo | NER Placebo/ASA Placebo
Diarrhea (Gastrointestinal disorders) | 2/91 | 7/90 | 5/90
Nausea (Gastrointestinal disorders) | 4/91 | 2/90 | 2/90
Vomiting (Gastrointestinal disorders) | 3/91 | 2/90 | 2/90
Fatigue (General disorders) | 1/91 | 2/90 | 0/90
Peripheral edema (General disorders) | 2/91 | 0/90 | 0/90
Sinusitis (Infections and infestations) | 1/91 | 2/90 | 1/90
Upper respiratory tract infection (Infections and infestations) | 3/91 | 2/90 | 2/90
Muscle strain (Injury, poisoning and procedural complications) | 2/91 | 1/90 | 0/90
Hyperglycemia (Metabolism and nutrition disorders) | 0/91 | 2/90 | 0/90
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/91 | 2/90 | 0/90
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2/91 | 0/90 | 0/90
Headache (Nervous system disorders) | 3/91 | 1/90 | 7/90
Insomnia (Psychiatric disorders) | 0/91 | 0/90 | 2/90
Urticaria (Skin and subcutaneous tissue disorders) | 2/91 | 1/90 | 0/90
Flushing (Vascular disorders) | 68/91 | 78/90 | 56/90
Hypertension (Vascular disorders) | 2/91 | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Provide ABBOTT at least sixty (60) days prior to submission for review, ABBOTT shall return comments within sixty (60) days of receipt of draft. Proposed draft shall be delayed an additional sixty (60) days in addition to the Review Period.